CLINICAL TRIAL: NCT06474416
Title: A Multicenter, Open-label, Single Dose, Phase Ⅰ Trial to Evaluate the Safety, Tolerability and Prelinminary Efficacy of BD111 in Patients With Herpes Simplex Virus Type I Stromal Keratitis in China
Brief Title: A Study of the Safety, Tolerability and Prelinminary Efficacy of BD111 in Herpes Simplex Virus Type I Stromal Keratitis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BD-HSK-111002-Ⅰ
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Herpes Simplex Virus Type I Stromal Keratitis
Keywords: Herpes simplex keratitis; Herpes Simplex Virus Type I; Stromal Keratitis
MeSH Terms: conditions — Keratitis, Herpetic | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- BD111 dose 1 group (Experimental): 1.25E+06 TU/eye
  Interventions: Genetic: BD111 Injection (Investigative New Drug)
- BD111 dose 2 group (Experimental): 2.5E+06 TU/eye
  Interventions: Genetic: BD111 Injection (Investigative New Drug)
- BD111 dose 3 group (Experimental): 5.0E+06TU/eye
  Interventions: Genetic: BD111 Injection (Investigative New Drug)
- BD111 dose 4 group (Experimental): 10E+06 TU/eye
  Interventions: Genetic: BD111 Injection (Investigative New Drug)
- Positive control group (Active Comparator): Triple-drugs therapy group: "Ganciclovir Eye gel+Valacilovir Tablets+Prednisolone Acetate Eye Drops" for 3 weeks.
  Interventions: Combination Product: Triple-drugs therapy of HSV-1 stromal keratitis

INTERVENTIONS:
Genetic: BD111 Injection (Investigative New Drug) — BD111 Injection (Investigative New Drug) is a type of lentiviral-like particle, which can simultaneously deliver SpCas9 and gRNA targeting the HSV-1 virus gene, also known as HSV-1-erasing lentiviral particles (HELP).
  Other Names: BD111 Lentivirus-like particles; HSV-1-erasing lentiviral particles; HELP
  Arms: BD111 dose 1 group; BD111 dose 2 group; BD111 dose 3 group; BD111 dose 4 group
Combination Product: Triple-drugs therapy of HSV-1 stromal keratitis — Triple-drugs therapy: "Ganciclovir Eye gel+Valacilovir Tablets+Prednisolone Acetate Eye Drops" for 3 weeks.
  Other Names: Ganciclovir Ophthalmic Gel; Valacyclovir Hydrochloride Tablets; Prednisolone Acetate Ophthalmic Suspension
  Arms: Positive control group

SUMMARY:
This Phase I study is intended to evaluate the safety, tolerability, PK/PD profiles and preliminary efficacy via corneal intrastromal administration in patients with herpes simplex virus-1 stromal keratitis (HSK), with a dose exploration of four ascending doses of BD111 (investigative drug product).

DETAILED DESCRIPTION:
Herpes simplex keratitis is an infectious diseases of the cornea that is primarily caused by Herpes Simplex Virus 1 (HSV-1). The stromal type, also known as HSV-1 stromal keratitis (HSK), is characterized by recurrent or chronic inflammation attributed to residual virus-triggered antigen-antibody-complement cascade reactions. BD111 is a lentivirus-like particle that is an active drug substance delivering gRNA-expressing cassettes and SpCas9 mRNA.The mechanism of action (MOA) is based on CRISPR/Cas9 gene editing technology.

This is a multicenter, open-label, dose-escalation, Phase I trial to evaluate the safety, tolerability, PK/PD profiles and preliminary efficacy of BD111 in patients with herpes simplex virus-1 stromal keratitis (HSK) in China. About 16 patients will be enrolled, dividing into open-label, four dose groups and one positive control (triple-drugs therapy) group. A rapid titration dose group combined with "3+3" dose escalation is designed for dose exploration.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the following inclusion criteria to be enrolled in this study

1. Aged 18 to 70 years old;
2. Clinically diagnosed patients with recurrent herpes simplex virus type I stromal keratitis (HSK). Definition of recurrence: the patient had been diagnosed with HSK and received "local antiviral eye drugs and oral antiviral drugs + local glucocorticoid eye drops" for 3 weeks with successful clinical efficacy. Before enrollment, the clinical recurrence of HSK occurred again with symptoms including tearing, photophobia, pain, blurred vision and foreign body sensation, and signs as recurrence of active inflammatory lesions examined by slit lamp;
3. HSV-1 nucleic acid test (qPCR method) positive;
4. No use of other systemic antiviral drugs or corticosteroids within 48 hours before enrollment;
5. No systemic immune diseases;
6. Good eyelid structure and blinking function;
7. Eye structure and function assessment showing potential for visual recovery;
8. No retinal detachment;
9. No history of corneal trauma;
10. The best visual acuity in the fellow eye (BCVA) ≥ 38 (ETDRS);
11. Fertile males or females must use highly effective contraceptive methods, such as, oral contraceptives, intrauterine devices, abstinence, or barrier contraception combined with spermicides, during the trial and continue contraception for 12 months after administration;
12. Participants voluntarily join the study, sign an informed consent form, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria: Patients with any of the following conditions cannot be enrolled in this study

1. Active ocular infection caused by other pathogens in the target eye or the fellow eye within 30 days before enrollment, including but not limited to infectious conjunctivitis, keratitis, scleritis, and endophthalmitis;
2. Patients with bilateral viral keratitis
3. Previous corneal transplant surgery in the study eye;
4. Any medicine or food allergic history;
5. Absence of tear film and blinking function;
6. Severe dry eye disease;
7. Ocular surface tumor;
8. Glaucoma;
9. Patients with systemic autoimmune diseases;
10. Signs of systemic infection before enrollment, including fever and receiving antibiotic treatment (systemic infection in this trial is defined as abnormal values in white blood cells, lymphocytes, and neutrophils in routine blood tests);
11. Severe diseases in the major organs including but not limited to cardiovascular, lung, liver, kidney, or other uncontrolled diseases;
12. HIV infection;
13. Pregnant and lactating women (pregnancy in this trial is defined as a positive urine or blood pregnancy test);
14. Participation in other drug or medical device clinical trials at present;
15. Alcohol or drug abuse;
16. Lack of compliance with the trial or the ability to sign an informed consent form;
17. Other situations deemed unsuitable for participation in the trial by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 12 months
  DLT is defined as toxicity related to BD111 observed by the investigator and sponsor during the treatment period, specifically: a) Endophthalmitis; b) Corneal perforation; c) Hypopyon; d) Other toxicities that are significantly worse than baseline or defined as ≥ Grade 4 ocular toxicity and persist for 14 days or longer, which require trial termination after discussion with the investigator and sponsor; e) Any non-ocular Grade ≥ 3 abnormality that persists for more than 1 week or requires hospitalization for medical intervention; f) death.
Maximum tolerated dose (MTD) | 12 months
  The highest dose at which ≤1/3 of the subjects experience DLT during the DLT observation period. The MTD dose must be confirmed in at least 6 subjects.
Recommended Phase 2 dose (RP2D) | 12 months
  The RP2D is determined by integrating safety, pharmacokinetic, and efficacy data from the comprehensive dose escalation. Typically, the MTD (DLT incidence ≤ 1/3) is used as the RP2D when it is confirmed, or a dose lower than the MTD is selected as the RP2D based on comprehensive data.
Incidence and characteristics of adverse events (AE) and serious adverse events (SAE) during the study | 12 months
  AE and SAE are recorded and evaluated, including eye-related AEs after treatment, such as AE at the corneal injection site.

SECONDARY OUTCOMES:
Tear fluid vector RNA | 12 months
  Tear fluid vector RNA copy numbers detected by real-time qPCR test, is one of Pharmacokinetics indicators of main components of BD111, and analysizing results will be used to evaluated the PK profile of tear fluid vector RNA and dose-response relationship of BD111.
Tear fluid vector circular DNA | 12 months
  Tear fluid vector circular DNA copy numbers detected by real-time qPCR test, is another Pharmacokinetics indicator of main components of BD111, and analysizing results will be used to evaluated the PK profile of tear fluid vector RNA and dose-response relationship of BD111.
Blood vector circular DNA | 12 months
  Real-time qPCR test will be used to detect copy number of vector circular DNA in blood, analysizing the PK profile of blood vector circular DNA and dose-response relationship of BD111.
Blood p24 protein | 12 months
  P24 protein concentration in blood will be assayed using ELISA p24 kit at preseted timepoints, analysizing the PK profile of Blood p24 protein.
Blood Cas9 protein | 12 months
  Cas9 protein concentration in blood will be assayed using ELISA p24 kit at preseted timepoints, analysizing the PK profile of Blood p24 protein.
Off-target Detection (Not applicable to comparison group) | 12 months
  BD111 off-target test of eye swabs samples will be conducted by DNA deep sequencing at Day 0, Day6 and Day 180 post-administration.
Antibodies to BD111-related ingredients (anti-drug antibodies, no applicable to comparison group) | 12 months
  Including: a) Anti-p24 antibody in the participants' blood samples at Day 0, Day 14, Day 28, Day 180 and Day 365; b) Anti-Cas9 antibody in the participants' blood samples at Day 0, Day 14, Day 28, Day 180 and Day 365; c) Anti-BD111 antibody in the participants' blood samples at Day 0, Day 14, Day 28, Day 180 and Day 365.
The percentage of participants with successful clearance of HSV-1 viral genome in tear at Day 14, Day 28, Day 70, Day 112, Day 180, and Day 365 post-administration | 12 months
  The definition of successful HSV-1 clearance: negative results in tear swab HSV-1 nucleic acid tests on two consecutive samplings (interval ≥14 days).
  The definition of a negative result in tear swab HSV-1 nucleic acid test: single qPCR Ct value = 40 or "undetected", or Ct value of the first qPCR test "36 < Ct value < 40", and the Ct value of repetitive qPCR test is 40 or "undetected".
The percentage of participants with failed clearance of HSV-1 viral genome in tears at Day 14, Day 28, Day 70, Day 112, Day 180, and Day 365 post-administration | 12 months
  The failure of HSV-1 viral genome clearance is determinated by HSV-1 positive results of qPCR test. HSV-1 positive definition of qPCR test: qPCR Ct value ≤ 36, or qPCR Ct value is "36 < Ct value < 40" and the Ct value of repetitive qPCR test is ≤ 36, or results of both qPCR tests are "36 < Ct value < 40".
Clinical cure rate of HSK at Day 70 and Day112 post-administration | 12 months
  Definition of HSK clinical cure: disappearance of the subject's clinical symptoms, disappearance of active inflammatory lesions on ophthalmologic examinations, and successful clearance of the HSV-1 viral genome.
The percentage of participants with HSK recurrence at Day 180, and Day 365 post-administration | 12 months
  Definition of HSK recurrence: HSV-1 nucleic acid qPCR test is positive, and clinical symptoms presents again, and ophthalmic examinations find active inflammatory lesions on interventional eye.
The score change of corneal inflammation scale post-administration | 12 months
  The score changes of corneal inflammation scale will be essessed at Day 70, Day 112, Day 180, and Day 365 post-administration.
The improvement in best corrected visual acuity (BCVA) | 12 months
  From baseline to Day 70, Day 112, Day 180, and Day 365 post-administration.
The improvement in corrected distance visual acuity (CDVA) post-administration | 12 months
  From baseline to Day 70, D11ay 2, Day 180, and Day 365 post-administration.

OTHER OUTCOMES:
Anti-p24 antibody in blood | 12 months
  At Day 14, Day 28, Day 180, and Day 365 post-administration.
Anti-Cas9 antibody in blood | 12 months
  At Day 14, Day 28, Day 180, and Day 365 post-administration.
Anti-BD111 antibody in blood | 12 months
  At Day 14, Day 28, Day 180, and Day 365 post-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, M.D., Principal Investigator — No. 270, West Academy Road, Wenzhou, Zhejiang, China
Locations (3):
- China (3):
  - Huashan Hospital, Fudan University, Shanghai, Shanghai City
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang